CLINICAL TRIAL: NCT01846494
Title: Longitudinal Assessment of Cardiovascular and Renal Health in Patients With Hepatitis-C (CARE-Hep C)
Acronym: CARE-Hep C
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00042419; Pro00044788 (Other: Duke eIRB Biorepository Protocol Number)
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2018-12

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Plasma, serum, and urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hepatitis C Virus (HCV) patients exposed to BMS-986094: Hepatitis C infected patients with previous exposure to BMS-986094
- HCV patients not exposed to BMS-986094: Hepatitis C patients without exposure to BMS-986094

SUMMARY:
The purpose of this study is to monitor the cardiovascular and renal health of patients who previously took BMS-986094 (an investigational medication for hepatitis C) in comparison to hepatitis C infected patients who have never taken BMS-986094.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be enrolled based on prior enrollment in the BMS 986094 studies or treatment-naïve HCV subjects with no known cardiovascular abnormalities.

1. All Subjects must give informed consent prior to participation in the study.
2. Subject participated in the Phase 1 or Phase 2 trials with BMS 986094 (including placebo arm) OR
3. Subject with known hepatitis C (Control)

   1. No previous exposure to BMS 986094
   2. Treatment naive at study entry (No prior hepatitis C treatment experience at the time of enrollment, including but not limited to: standard interferon, pegylated interferon, ribavirin, boceprevir, telaprevir, or other experimental drugs for hepatitis C).

Exclusion Criteria

1. For subjects who participated in the Phase 1 or Phase 2 trials with BMS 986094, there are no exclusion criteria
2. For the control group of subjects without exposure to BMS 986094, the following exclusion criteria, based on clinically available data, apply:

   1. Signs or symptoms of decompensated liver disease such as variceal bleeding, ascites, hepatic encephalopathy, active jaundice defined by an indirect bilirubin >2, ALT or AST laboratory values ≥ 10 times the upper limit of normal, or other evidence of decompensated liver disease or hepatocellular carcinoma
   2. Chronic liver disease other than HCV not limited to Hepatitis B virus (positive test for HBsAg), hemochromatosis, auto-immune hepatitis, alcoholic liver disease or non-alcoholic fatty liver disease
   3. History of liver transplantation
   4. Co-infection with HIV (positive test for anti-HIV Ab)
   5. Prior history of cardiomyopathy (ejection fraction ≤ 50%) or history of heart failure
   6. Signs or symptoms of decompensated heart failure or
   7. Prior history of coronary artery disease, acute myocardial infarction or coronary artery revascularization (percutaneous or coronary artery bypass grafting)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hepatitis C positive subjects previously exposed to BMS 986094 and Hepatitis C positive subjects not previously exposed to BMS 986094.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2013-05-10 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian F. Hernandez, MD, Principal Investigator — Duke Clinical Research Institute
Locations (13):
- United States (12):
  - Anaheim Clinical Trials, Anaheim, California
  - Scripps Clinic, San Diego, California
  - Tuan Nguyen, MD, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Kansas City Gastroenterology and Hepatology, Kansas City, Missouri
  - Weill Cornell Medical Center, New York, New York
  - Asheville Gastroenterology Associates, PA, Asheville, North Carolina
  - Options Health Research, Tulsa, Oklahoma
  - Lancaster Heart Foundation, Lancaster, Pennsylvania
  - Central Texas Clinical Research, Austin, Texas
  - Alamo Medical Research, San Antonio, Texas
- Fundacion de Investigation de Diego, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 113 participants recruited from 10 May 2013 (first participant first visit) to 10 Mar 2018 (last participant last visit) at 15 clinical sites. One participant was followed by the Duke Clinical Research Institute (DCRI) call center.
Period: Overall Study
Arm/Group | HCV Patients Not Exposed to BMS-986094 | Hepatitis C Virus (HCV) Patients Exposed to BMS-986094
Started | 50 | 63
Completed | 20 | 25
Not Completed | 30 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HCV Patients Not Exposed to BMS-986094 | Hepatitis C Virus (HCV) Patients Exposed to BMS-986094 | Total
Number analyzed (Participants) | 50 | 63 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (9.74) | 50.2 (9.74) | 51.9 (9.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 30 | 41 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 13 | 28
  Not Hispanic or Latino | 35 | 50 | 85
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 2 | 11
  White | 38 | 57 | 95
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Death or Rehospitalization Due to Cardiovascular or Renal Cause
Time Frame: 5 years
Population: Only subjects who were assessed at least once for each component of the composite endpoint were included for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | HCV Patients Not Exposed to BMS-986094 | Hepatitis C Virus (HCV) Patients Exposed to BMS-986094
Number analyzed (Participants) | 46 | 57
Participants | 1 | 2

2. Secondary Outcome: Composite of Death and Cardiovascular and Renal Dysfunction
Description: Reported as percentage of participants experiencing one or more of the following endpoints: all-cause mortality, rehospitalization for cardiac/renal cause, increase in BNP to >100 or doubling from baseline, new onset of LVEF <50%, new onset of eGFR <60% or >= 25% reduction from baseline.
Time Frame: 5 years
Measure: Number; unit: percentage of participants
Arm/Group | HCV Patients Not Exposed to BMS-986094 | Hepatitis C Virus (HCV) Patients Exposed to BMS-986094
Number analyzed (Participants) | 50 | 63
percentage of participants | 31.1 | 35.2
Statistical Analysis 1: Comparison: HCV Patients Not Exposed to BMS-986094 vs Hepatitis C Virus (HCV) Patients Exposed to BMS-986094; Test type: Other; p = 0.6173, Log Rank

ADVERSE EVENTS:
Time Frame: 58 months
Description: Non-serious adverse events were not collected. Collection, evaluation, and reporting of serious adverse events (SAEs) was limited to SAEs related to cardiac and renal events dysfunction and SAEs resulting in death. Serious adverse events were collected and recorded on the SAE page of the eCRF from the signing of informed consent to the end of the follow-up period.
Arm/Group | HCV Patients Not Exposed to BMS-986094 | Hepatitis C Virus (HCV) Patients Exposed to BMS-986094
All-Cause Mortality (participants affected / at risk) | 1/50 | 2/63
Serious Adverse Events (participants affected / at risk) | 1/50 | 2/63
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HCV Patients Not Exposed to BMS-986094 (N=50) | Hepatitis C Virus (HCV) Patients Exposed to BMS-986094 (N=63)
Death (General disorders) | 1 | 0 — Not attributed to cardiac or renal dysfunction.
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT01846494/Prot_SAP_000.pdf